CLINICAL TRIAL: NCT02351284
Title: Impact of Hypovitaminosis D in Metabolic Disturbances and Bone Metabolism, and Changes in Patients Receiving Vitamin D Supplementation
Brief Title: Impact of Hypovitaminosis D on Bone Disease in HIV Infected Patients
Acronym: PuraVIHta
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jose L. Casado (Network)
Responsible Party: Sponsor-Investigator, Jose L. Casado, MD, PhD, Asociacion para el Estudio de las Enfermedades Infecciosas
Organization: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Other Study IDs: 20/15
Record Dates: First submitted 2015-01-23; First posted 2015-01-30 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Hypovitaminosis D
Keywords: HIV, vitamin D, osteoporosis
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measurement — Measurement of vitamin D, PTH, and BMD changes in HIV-infected patients

SUMMARY:
To determine the prevalence of hypovitaminosis D in HIV infected patients, and the consequences on secondary hyperparathyroidism, and bone mineral density (BMD). Also, to establish the improvement in vitamin D status, parathyroid hormone (PTH) and BMD, in case of receiving vitamin D supplementation, during a follow up period of at least 1 year.

DETAILED DESCRIPTION:
This study deals with the impact of vitamin D on metabolism and bone health in HIV infected patients. To answer the questions about the importance of this hormone in this population, we designed a cohort study about the prevalence of vitamin D deficiency (measured as 25-hydroxy-vitamin D), classifying it in severe deficiency (<10 ng/ml), deficiency (< 20 ng/ml), or insufficiency (< 30 ng/ml), the relationship with secondary hyperparathyroidism (PTH > 65 pg/ml), and related BMD by dual X-ray absorptiometry (DXA). These results will be adjusted by baseline factors, such as age, gender, body mass index (BMI), hepatitis C virus (HCV) coinfection, risk practice for HIV infection, CD4+ count, antiretroviral therapy, and HIV RNA level.

In patients receiving vitamin D supplementation according to clinical decision, it will be evaluated the changes in percentage of hypovitaminosis D and/or secondary hyperparathyroidism, and the effect on BMD. Bone biomarkers will be collected to determine the impact of changes secondary to vitamin D improvement in the bone evolution.

ELIGIBILITY:
Inclusion Criteria:

* HIV older than 18 years

Exclusion Criteria:

* Chronic kidney disease stage 4 and 5 (creatinine clearance < 30 ml/min)
* Pregnancy
* Uso of corticosteroid therapy, or requiring anti-resorptive treatment
* Prolonged hospitalization or internment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients in follow up
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of osteopenia/osteoporosis and secondary hyperparathyroidism in HIV infected patients according to vitamin D strata | 48 weeks
  Percentage of patients with high PTH and reduced BMD in each vitamin D strata (< 10 ng/ml, 10-20 ng/ml, 20-30 ng/ml, > 30 ng/ml)

SECONDARY OUTCOMES:
Changes in vitamin D levels secondary to seasonality | 48 weeks
  Changes in 25-hydroxy vitamin D according to season
Efficacy of supplementation in reducing secondary hyperparathyroidism and osteopenia/osteoporosis | 48 weeks
  Changes in PTH and BMD (% of patients having secondary hyperparathyroidism and osteopenia/osteoporosis) after receiving vitamin D supplementation according to clinical decision
Impact of vitamin D levels (25OHD) in reducing phosphaturia levels | 48 weeks
  Improvement in phosphaturia levels (elemental urine) according to vitamin D strata and/or supplementation
Correlation between values of bone biomarkers (osteocalcin, beta-crosslaps, alkaline phosphatase, P1NP) and rates of osteopenia/osteoporosis | 48 weeks
  To establish baseline values and relationship of bone biomarkers with bone mineral density status, adjusted by vitamin D strata

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bañon, MD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain